CLINICAL TRIAL: NCT04792125
Title: The Effects of External Electrical Stimulation Added to Pelvic Floor Muscle Training in Women With Stress Incontinence
Brief Title: Effect of External Electrical Stimulation and Pelvic Floor Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Ulkukezbansahin, PhD, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-55
Record Dates: First submitted 2021-02-28; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Urinary Incontinence, Stress; Electrical Stimulation; Pelvic Floor Disorders; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- External electrical stimulation (EES) added to pelvic floor muscle training (PFMT) group (Experimental): This arm is going to include the patients who are performed external electrical stimulation (EES) added to pelvic floor muscle training (PFMT).
  Interventions: Behavioral: External electrical stimulation (EES) added to pelvic floor muscle training (PFMT)
- External electrical stimulation (EES) group (Other): This arm is going to include the patients who are performed external electrical stimulation (EES).
  Interventions: Behavioral: External electrical stimulation
- Pelvic floor muscle training (PFMT) group (Active Comparator): This arm is going to include the patients who are performed pelvic floor muscle training (PFMT).
  Interventions: Behavioral: Pelvic floor muscle training (PFMT)

INTERVENTIONS:
Behavioral: External electrical stimulation (EES) added to pelvic floor muscle training (PFMT) — Patients will be treated with the Innovo device using eight external electrodes with a combined stimulator. Electrodes will be applied to the buttocks, outer hips and anterior and posterior proximal thighs 3 days a week for 30 minutes each session.
  While explaining the exercise to the patients, it was stated that 1 set of exercise consisted of 10 fast contractions and 10 slow contractions. For the first 2 weeks, they were asked to exercise 2 sets a day, every day. Thus, in the first 2 weeks, 20 fast contractions and 20 slow contractions were performed. Then, 2 sets were increased every two weeks and the exercise was ended as 8 sets (80 fast and 80 slow contractions) at the end of the 8th week.
  Arms: External electrical stimulation (EES) added to pelvic floor muscle training (PFMT) group
Behavioral: External electrical stimulation — Patients will be treated with the Innovo device using eight external electrodes with a combined stimulator. Electrodes will be applied to the buttocks, outer hips and anterior and posterior proximal thighs 3 days a week for 30 minutes each session.
  Arms: External electrical stimulation (EES) group
Behavioral: Pelvic floor muscle training (PFMT) — While explaining the exercise to the patients, it was stated that 1 set of exercise consisted of 10 fast contractions and 10 slow contractions. For the first 2 weeks, they were asked to exercise 2 sets a day, every day. Thus, in the first 2 weeks, 20 fast contractions and 20 slow contractions were performed. Then, 2 sets were increased every two weeks and the exercise was ended as 8 sets (80 fast and 80 slow contractions) at the end of the 8th week.
  Arms: Pelvic floor muscle training (PFMT) group

SUMMARY:
In this study, the effects of the external electrical stimulation (EES) added to pelvic floor muscle training (PFMT) on stress urinary incontinence (SUI) were investigated.

DETAILED DESCRIPTION:
Fifty one women with mild and moderate SUI symptoms were included in the study. The patients were divided into three groups of PFMT (n:17), EES (n:17) and PFMT+ EES (n:17) by block randomization. The PFMT was applied every day of the week, and EES was applied 3 days a week for 8 weeks. Pelvic floor muscle strength (PFMS), pelvic floor muscle endurance, subjective perception of improvement, severity of incontinence, quality of life, pelvic floor dysfunction (PTD) and urinary parameters were assessed as outcome variables. All measurements, except subjective perception of improvement were investigated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* having symptoms of pure stress urinary incontinence and stress predominant UI
* ability to contract pelvic floor muscle strength
* Having a mild or moderate SUI symptom according to the 24-hour pad test results.

Exclusion Criteria:

* Pregnancy,
* Having been treated for incontinence within a period of six months ago,
* Not being able to cooperate,
* Presence of urinary infection
* Use of metal implants or cardiac pacemakers,
* Epilepsy,
* Presence of stage 3 or 4 pelvic organ prolapse,
* Presence of accompanying neurological disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Self-reported improvement | 8 weeks
  Perception of urinary incontinence improvement compared with baseline was assessed using four-item Likert-type scale (worse, same, better, cured).

SECONDARY OUTCOMES:
24 hour pad test | 8 weeks
  Urinary incontinence severity was assessed.
pelvic floor muscle strength and endurance | 8 weeks
  measured using noninvasive vaginal perineometer

CONTACTS AND LOCATIONS:
Overall Officials: ULKU K SAHIN, PhD, Principal Investigator — Giresun University
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Kaya S, Akbayrak T, Gursen C, Beksac S. Short-term effect of adding pelvic floor muscle training to bladder training for female urinary incontinence: a randomized controlled trial. Int Urogynecol J. 2015 Feb;26(2):285-93. doi: 10.1007/s00192-014-2517-4. Epub 2014 Sep 30. PMID 25266357
- [Result] Turkan A, Inci Y, Fazli D. The short-term effects of physical therapy in different intensities of urodynamic stress incontinence. Gynecol Obstet Invest. 2005;59(1):43-8. doi: 10.1159/000081133. Epub 2004 Sep 29. PMID 15459518
- [Result] Huebner M, Riegel K, Hinninghofen H, Wallwiener D, Tunn R, Reisenauer C. Pelvic floor muscle training for stress urinary incontinence: a randomized, controlled trial comparing different conservative therapies. Physiother Res Int. 2011 Sep;16(3):133-40. doi: 10.1002/pri.489. Epub 2010 Sep 16. PMID 20848671
- Available data/document: Study Protocol: 31270846 — https://pubmed.ncbi.nlm.nih.gov/31270846/ — External electrical stimulation compared with intravaginal electrical stimulation for the treatment of stress urinary incontinence in women: A randomized controlled noninferiority trial